CLINICAL TRIAL: NCT00780039
Title: Phase II, Open-Label, Study of CAELYX and Carboplatin Intermediate Platinum-Sensitive (6-12 Months Treatment-free Interval) Relapsed Epithelial Ovarian Cancer.
Brief Title: A Study to Evaluate the Safety and Efficacy of Caelyx in Combination With Carboplatin in Patients With Ovarian Cancer Recurrent Within Six to Twelve Months After Initial Carboplatin and Paclitaxel Chemotherapy (P03625)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03625
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Caelyx 30 mg/m2 in combination with carboplatin dosed to target AUC of 5 mg/mL.min.
  Interventions: Drug: Pegylated Liposomal Doxorubicin; Drug: Carboplatin

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin — Subjects will receive Caleyx 30 mg/m2 intravenously on Day 1 of each 4-week cycle, during 6 cycles. Patients still achieving clinical benefit after a total of 6 cycles may continue therapy.
  Other Names: SCH 200746
Drug: Carboplatin — Subjects will receive carboplatin dosed to target AUC of 5 mg/mL.min, intravenously, on Day 1 of each 4-week cycle, after the Caelyx infusion, during 6 cycles. Patients still achieving clinical benefit after a total of 6 cycles may continue therapy.

SUMMARY:
Doxorubicin has been used to treat ovarian cancer as part of different combination therapies, but high cumulative doses should be avoided because of the risk of cardiotoxicity. Pegylated Liposomal Doxorubicin (Caelyx) has been developed to reduce the risk of cardiotoxicity. The purpose of this study is to evaluate the safety and efficacy of Caelyx in combination with carboplatin in women with recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* Subject must have histological diagnosis of epithelial ovarian cancer
* Subject must have received a taxane and platinum regimen and have maintained a treatment-free status for at least six months and not more than twelve months following completion of first line therapy.
* Subject must have measurable ovarian cancer by appropriate radiological imaging.
* ECOG performance Score of 0 or 1.
* Subject's life expectancy must be > 6 months.
* Subject must have normal organ function, except if abnormal due to tumor involvement:

  * Adequate bone marrow function (platelets >=100 X 10^9/L, hemoglobin >=100 g/L, neutrophils >=1.5 X 10^9/L)
  * Adequate renal function (serum creatinine<=1.5 X the upper limit of normal (ULN)
  * Adequate liver function (bilirubin and AST or ALT<=2 times ULN, unless related to primary disease.
* MUGA scan must indicate left ventricular ejection fraction above 90%.
* Women of childbearing potential must be using adequate contraception (prescribed under medical supervision) and have a negative pregnancy test at the time of enrollment.
* Subject must be able to sign written informed consent.

Exclusion Criteria:

* Subject who is pregnant or is breast feeding.
* Subject who has history of cardiac disease, with New York Heart Association Class II or greater.
* Subject with a history of severe hypersensitivity reactions to products containing Cremophor® EL.
* Subject with clinically significant hepatic disease.
* Subject who has uncontrolled bacterial, viral, or fungal infection.
* Subject who exhibits confusion or disorientation.
* Subject with any condition that would prevent adequate follow-up.
* Subject with a history of prior malignancy treated with systemic chemotherapy or radiotherapy.
* Subject who has received two or more prior chemotherapy regimens for ovarian cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2007-09-06 (Actual); Study Completion 2007-09-06 (Actual)

PRIMARY OUTCOMES:
Complete response rate, according to RECIST criteria; Partial response rate, according to RECIST criteria | Complete or partial response: re-evaluation 4 weeks later to confirm response; Upon completion of chemotherapy: follow-up every 2 months until documentation of progressive disease; All patients will be followed for a minimum of one year for survival

SECONDARY OUTCOMES:
Safety and tolerability; Duration of response; CA-125 response; Time to progression; Overall survival | All patients will be followed for a minimum of one year for survival

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Li KJ, Garoff H. Packaging of intron-containing genes into retrovirus vectors by alphavirus vectors. Proc Natl Acad Sci U S A. 1998 Mar 31;95(7):3650-4. doi: 10.1073/pnas.95.7.3650. PMID 9520420
- [Derived] Power P, Stuart G, Oza A, Provencher D, Bentley JR, Miller WH Jr, Pouliot JF. Efficacy of pegylated liposomal doxorubicin (PLD) plus carboplatin in ovarian cancer patients who recur within six to twelve months: a phase II study. Gynecol Oncol. 2009 Sep;114(3):410-4. doi: 10.1016/j.ygyno.2009.04.037. Epub 2009 Jun 10. PMID 19520420